CLINICAL TRIAL: NCT05303259
Title: Effect of Bevacizumab on Asymptomatic Radiotherapy-induced Brain Injury in Patients With Head and Neck Cancer
Brief Title: Effect of Bevacizumab on Asymptomatic Radiotherapy-induced Brain Injury
Acronym: BRAIN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-KY-095
Record Dates: First submitted 2021-12-19; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-07

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HNC patients with radiation-induced brain injury. (Experimental): Bevacizumab 2.5mg/kg， q2w，4 cycles.
  Interventions: Drug: Bevacizumab
- HNC patients without brain injury after radiotherapy. (No Intervention): No treatment.

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 2.5mg/kg, q2w, 4 cycles.
  Arms: HNC patients with radiation-induced brain injury.

SUMMARY:
To investigate the effect of Bevacizumab on asymptomatic radiotherapy-induced brain injury patients with head and neck cancer.

DETAILED DESCRIPTION:
Radiotherapy-induced brain injury (RI) is a serious complication of radiotherapy in head and neck cancer (HNC) patients. Previous studies have confirmed that Bevacizumab has a good effect on patients with symptomatic RI .However, patients with RI maybe do not show clinical symptoms in the early stage. The clinical symptoms will appear with the progression of the RI lesion. There has been no relevant research on whether early intervention is necessary for asymptomatic RI. The investigators conduct this multicenter, randomized clinical research to explore the efficacy and safety of Bevacizumab in asymptomatic RI.

ELIGIBILITY:
Inclusion Criteria:

Head MRI confirmed RI lesions. Sign the informed consent.

Exclusion Criteria:

With clinical symptoms of RI lesions. Head MRI showed bleeding lesions Contraindications of Bevacizumab. Pregnant women and parturient women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and duration of onset of clinical symptoms. | Change form baseline to evaluation at 1 year.
  The incidence and duration of onset of clinical symptoms within 1 year after treatment between the treatment group and the control group.

SECONDARY OUTCOMES:
change of RI volume. | Change form baseline to evaluation at 1 year.
  The change of RI volume between the treatment group and the control group.
change of cognitive function. | Change form baseline to evaluation at 1 year.
  The change of cognitive function (MoCa scores) between the treatment group and the control group. The MoCA score ranges from 0 to 30, and higher scores mean a better outcome.
overall survival | Change form baseline to evaluation at 1 year.
  the overall survival between the treatment group and the control group.
change of quality of life. | Change form baseline to evaluation at 1 year.
  The change of quality of life ( WHOQOL scale) between the treatment group and the control group. The higher the QOL scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Ph.D, Study Chair — sun yat-sen memorial hospital,sun yat-sen universicy
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No